CLINICAL TRIAL: NCT03726619
Title: e-CHEC-uP: Scaling up an Efficacious Cancer Screening Intervention for Women With Limited English
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IRB00180383
Record Dates: First submitted 2018-10-30; First posted 2018-10-31 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer; Cervical Cancer
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-CHEC-uP (Experimental): Group 1 will receive the education study intervention after the first baseline questionnaire. Participants will be asked to take part in a one-time, 1 to 1.5-hour online education on breast and cervical cancer prevention followed by monthly phone calls and navigation assistance by a community health worker to help address any barriers in order to help receive a mammogram or a Pap test.
  Interventions: Behavioral: e-CHEC-uP
- CHEC-uP (Active Comparator): Group 2 will receive a similar education intervention but the education is offered face-to-face instead. Participants will be asked to take part in a one-time, 1 to 1.5-hour face-to-face education on breast and cervical cancer prevention followed by monthly phone calls and navigation assistance by a community health worker.
  Interventions: Behavioral: CHEC-uP

INTERVENTIONS:
Behavioral: e-CHEC-uP — One time online-based education about breast and cervical cancer screening procedures followed by phone counseling by trained community health worker over 6 months
  Arms: e-CHEC-uP
Behavioral: CHEC-uP — One time face-to-face education about breast and cervical cancer screening procedures followed by phone counseling by trained community health worker over 6 months
  Arms: CHEC-uP

SUMMARY:
This research is being done to learn more about whether or not Korean American women will improve the screening practices for breast and cervical cancer if subjects receive education and follow-up from community health workers. The education materials may be given via online or in-person. Primary Hypothesis: e-CHEC-uP will be as efficacious as the original CHEC-uP in promoting mammogram and Pap test screening among Korean immigrant women (KIW) at 6 months.

Objectives: (1) To develop a web-based platform of the health literacy education component of the original CHEC-uP intervention; (2) To evaluate the acceptability and usability of the web version of the health literacy education in a user testing sample of 10 KIW; and (3) To conduct a pilot study to test the preliminary efficacy of the web version of CHEC-uP (e-CHEC-uP) in 40 KIW.

DETAILED DESCRIPTION:
e-CHEC-uP stands for e-Community based breast and cervical cancer control education program.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65 years
* Self-identified as a Korean American woman
* Overdue for a mammogram (40-65 years of age only) or a Pap test**
* Able to read and write Korean or English
* Willing to provide written consent to allow the researchers to audit medical records for mammography and Pap test use

Exclusion Criteria:

* A cancer diagnosis
* Being pregnant
* An acute and/or terminal condition (e.g., life expectancy of less than 6 months or last cancer treatment within the last 5 years)
* Psychiatric diagnosis (e.g., schizophrenia or cognitive impairment) or other conditions that preclude participation in the study activities
* Had undergone a hysterectomy

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — self-identified as a Korean American woman
Enrollment: 40 (Actual)
Dates: Start 2019-07-14 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Age-appropriate mammogram screening test | 6 months
  Patient medical records will be reviewed to confirm the receipt of mammogram and whether the age at which it was received is "appropriate". According to the American Cancer Society (ACS), Mammograms received from ages 40 to 54 years (annual screening) and from ages 55 years onward (biennial screening) will be deemed appropriate. It is optional to continue annual screening after age 54 years based on a woman's choice.
  The investigators will compare the proportion of women in each group (e-CHEC-uP intervention vs. CHEC-uP) who completed mammogram at 6 months.
Age-appropriate Pap screening test | 6 months
  Patient medical records will be reviewed to confirm the receipt of Pap test and whether the age at which it was received is "appropriate". According to the American Cancer Society (ACS), Pap tests received from ages 21 to 65 years once every 3 years will be deemed appropriate.
  The investigators will compare the proportion of women in each group (e-CHEC-uP intervention vs. CHEC-uP) who completed Pap test at 6 months.

SECONDARY OUTCOMES:
Health Literacy as assessed by a 49-item instrument | 6 months
  Scoring of the health literacy instrument is in such a way that each correct response will be coded as 1 whereas incorrect response will be coded as 0. Total scores can range from 0 to 49 with higher scores indicating higher health literacy.
Breast Cancer knowledge as assessed by a 25-item instrument | 6 months
  Scoring of the breast cancer knowledge instrument is in such a way that each correct response will be coded as 1 whereas incorrect response will be coded as 0. Total scores for breast cancer knowledge will range from 0 to 25. Higher scores indicate higher breast cancer knowledge.
Cervical Cancer knowledge as assessed by 10-item instrument | 6 months
  Scoring of the cervical cancer knowledge instrument is in such a way that each correct response will be coded as 1 whereas incorrect response will be coded as 0. Total scores for cervical cancer knowledge will range from 0 to 10. Higher scores indicate higher cervical cancer knowledge.
Cancer screening-related self-efficacy as assessed by 8-item scale | 6 months
  Scoring of the cancer screening-related self-efficacy is to assess one's belief about ability to get cancer screening. The 8-item scale (developed by the study team) scoring ranges from "not at all confident" coded as 1 to "very confident" coded as 4 for each item. Total scores will range from 8 to 32 with higher scores indicating higher self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Hae-Ra Han, PhD, RN, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Han HR, Huh B, Kim MT, Kim J, Nguyen T. Development and validation of the assessment of health literacy in breast and cervical cancer screening. J Health Commun. 2014;19 Suppl 2(0 2):267-84. doi: 10.1080/10810730.2014.936569. PMID 25315598
- [Background] Park S, Chang S, Chung C. Effects of a cognition-emotion focused program to increase public participation in Papanicolaou smear screening. Public Health Nurs. 2005 Jul-Aug;22(4):289-98. doi: 10.1111/j.0737-1209.2005.220404.x. PMID 16150010
- [Background] McCance KL, Mooney KH, Smith KR, Field R. Validity and reliability of a breast cancer knowledge test. Am J Prev Med. 1990 Mar-Apr;6(2):93-8. PMID 2363955
- [Derived] Hwang DA, Lee A, Song JM, Han HR. Recruitment and Retention Strategies Among Racial and Ethnic Minorities in Web-Based Intervention Trials: Retrospective Qualitative Analysis. J Med Internet Res. 2021 Jul 12;23(7):e23959. doi: 10.2196/23959. PMID 34255658